CLINICAL TRIAL: NCT02974959
Title: Vagus Nerve Stimulation to Treat Mild To Moderate Traumatic Brain Injury
Brief Title: Vagus Nerve Stimulation to Treat Moderate Traumatic Brain Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CentraCare (Other)
Collaborators: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSR 16-4171
Record Dates: First submitted 2016-09-12; First posted 2016-11-29 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Traumatic Brain Injury; Acute Brain Injuries
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the study coordinator had access to the master list which noted whether the device was active or a sham. This information was not provided to or accessible by the participants, care providers, investigators, or outcome assessors.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gammaCore active device (Experimental): Patients in this arm will be using an active device which delivers a treatment dose of current to the vagus nerve twice daily for 120 seconds
  Interventions: Device: gammaCore active device
- gammaCore Sham device (Sham Comparator): Patients in this arm will be using a sham device which does not deliver a treatment dose of current, but will deliver enough current to cause tingling on the skin.
  Interventions: Device: gammaCore sham device

INTERVENTIONS:
Device: gammaCore active device — The nVNS therapy will be performed using the gammaCore-R (electroCore LLC, NJ), which is an external hand-held vagal nerve stimulator. The gammaCore-R produces a low voltage electric signal consisting of five 5000 Hz pulses that are repeated at a rate of 25 Hz. It allows for a 120 second stimulation session. The stimulation will occur twice daily, one time in the morning and one time in the evening. This should be done as close to 12 hours apart as possible and should occur twice daily for the entire 12 week study period.
  Arms: gammaCore active device
Device: gammaCore sham device — The sham device appears identical to the gammaCore but does not provide a frequency of stimulation powerful enough to stimulate either efferent or afferent fibers of the vagus nerve. However, it does supply a low frequency current which will cause a tingling of this skin to improve blinding of the patients.
  Arms: gammaCore Sham device

SUMMARY:
The purpose of this single-center, prospective, randomized (1:1), double-blind, sham-controlled parallel-arm pilot study is to provide initial evidence of use of the noninvasive vagus nerve stimulator for treatment in patients recovering from concussion and moderate traumatic brain injury to improve clinical recovery. The study compares the safety and effectiveness of an active gammaCore treatment against a sham treatment.

DETAILED DESCRIPTION:
Our primary aim is to assess for evidence of the effectiveness of the nVNS in reducing clinical symptoms such as motor and cognition deficits. As a primary endpoint, we will analyze the difference between groups at all time points in standardized cognitive assessments. We will also assess the levels of different inflammatory cytokines.

The secondary endpoints for moderate TBI are functional assessments and quality of life questionnaires including a depression screen. Our secondary aim is to assess the safety of a non-invasive VNS (nVNS) in a subset of patients who have suffered a moderate TBI. We do not anticipate any significant difference between heart rate variability (HRV) in active compared to sham treatments and no difference symptoms experienced during treatment sessions.

We propose a single-center, prospective, randomized (1:1), double-blind, sham-controlled, parallel-arm pilot study. We determined that an N of 30 patients would be needed to reach significance. Moderate TBI will be defined by the Head Injury Interdisciplinary Special Interest Group of the American Congress of Rehabilitation Medicine (full list in inclusion criteria) seeking care at HCMC within 2 weeks of injury. Recruited subjects will be randomized to active treatment or sham-treatment control arms. Randomization to active or sham gammaCore treatment will occur during the screening visit after enrollment, and intervention will begin at the baseline visit that occurs 72 hours (+/- 1 day) after enrollment. Informed consent will be obtained from patients or their proxy prior to enrollment. If a proxy elects to enroll a patient, who then recovers during the course of the study, they will be able to withdraw from the study if they so desire. We anticipate enrollment to take approximately 6 months, and enrolled subjects will be followed through the final week 18 follow up visit, estimating a completion date 9 months after the first enrollment.

The treatment will include 12 weeks of active interventional therapy, with seven visits, including the screening visit that takes place within 2 weeks of injury. From the baseline visit, there will be a follow up phone call at 1 week, and a follow up visit at 2, 6, 12 and 18 weeks. During each of these visits, data assessing heart rate variability will be obtained using a chest strap heart rate monitor and a non-invasive heart rate variability monitor will be used to measure minute phenomenon in heartbeats. This will be done while supine, during treatment and after an orthostatic challenge (i.e. standing or sitting upright). An EKG will be obtained at each visit to assess for bradycardia.

The nVNS therapy will be performed using the gammaCore-R (electroCore LLC, NJ), which is an external hand-held vagal nerve stimulator. The gammaCore-R produces a low voltage electric signal consisting of five 5000 Hz pulses that are repeated at a rate of 25 Hz. The strength of the stimulation is lower than that required to activate efferent vagal nerve fibers that mediates cardiac specific effects and will only be used on the left vagus nerve, which has fewer cardiac projections. It allows for a 120 second stimulation session. The stimulation will occur twice daily, one time in the morning and one time in the evening. This should be done as close to 12 hours apart as possible and should occur twice daily for the entire 12 week study period. The sham device appears identical to the gammaCore but does not provide a frequency of stimulation powerful enough to stimulate either efferent or afferent fibers of the vagus nerve. However, it does supply a low frequency current which will cause a tingling of this skin to improve blinding of the patients. After the 12 week visit, the device will be returned. However, both the treating physician and the patient will remain blinded to the study arms until the completion of the study at week 18. Blood samples (10 mL or two teaspoons) will be drawn at the screening visit, as well as the 12 and 18-week time points for biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent obtained by Subject or Subject's proxy.
2. Is between the ages of 18 and 60 years, male or female.
3. Meets the criteria of the Head Injury Interdisciplinary Special Interest Group of the American Congress of Rehabilitation Medicine, which defines a head injury as a traumatically induced physiologic disruption of brain function, as manifested by one of the following:

   * Any period of loss of consciousness (LOC),
   * Any loss of memory for events immediately before or after the accident,
   * Any alteration in mental state at the time of the accident,
   * Focal neurologic deficits, which may or may not be transient.
4. Meets the criteria for moderate TBI as defined by the Head Injury Interdisciplinary Special Interest Group of the American Congress of Rehabilitation Medicine, which are as follows:

   * Length of stay at least 48 hours,
   * Glasgow Coma Scale (GCS score of 9-12 or higher)
   * Operative intracranial lesion,
   * Abnormal CT scan findings.
5. Has had a craniotomy, but those with hydrocephalus or active intracranial pressure elevation will be excluded.
6. Able to accurately communicate the sensation of amplitude of intensity by the stimulation treatment with the GammaCore device.
7. Has a stable orthopedic or other traumatic body injury.
8. Is capable of completing all study assessments.
9. Agrees to use the GammaCore device as intended and follow all of the requirements of the study, including follow-up visits.
10. Agrees to record usage of the GammaCore device, all required study data, and report any adverse effects to the sponsor/investigator within 24 hours of any such adverse event.

Exclusion Criteria:

1. Has an active DNR/DNI (do not resuscitate/ do not intubate) request.
2. Has dissent among family members / next of kin regarding level of care.
3. Has a penetrating injury.
4. Has concurrent active severe medical problems or conditions, which could prevent survival during the course of the study.
5. Has pre-existing central nervous system disease or associated comorbidities that may not allow for an 18-week follow-up visit.
6. Has an abscess, infection or lesion (including lymphadenopathy) at the gammaCore treatment site.
7. Has known or suspected moderate to severe atherosclerotic cardiovascular disease, carotid artery disease (e.g. bruits or history of TIA or CVA).
8. Has a clinically significant irregular heart rate or rhythm.
9. Has uncontrolled hypertension (systolic bp > 200 or diastolic bp >100), recent (within the last 3 months) heart attack, recent (within the last 3 months) stroke, known aortic aneurysm, or congestive heart failure (CHF).
10. Is currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker, defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant.
11. Has a history of significant carotid endarterectomy, vagotomy, dysaesthesia or vascular neck surgery on either side of the neck.
12. Has been implanted with metal cervical spine hardware.
13. Has a recent or repeated history of syncope.
14. Has a recent or repeated history of seizures.
15. Has known clotting disorder or hemophilia
16. Has anemia (hb<12)
17. Is pregnant or nursing, or of childbearing potential and is unwilling to use an accepted form of birth control (hormonal, barrier method, surgical, or abstention or is at least two years post-menopause).
18. Is participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days.
19. Is an employee of the clinical study site or a relative of the Investigator.
20. Has an abnormal baseline electrocardiogram (ECG), including second and third degree heart block, atrial fibrillation, atrial flutter, recent history of ventricular tachycardia or ventricular fibrillation or clinically significant premature ventricular contraction.
21. Has a known history or suspicion of substance abuse or addiction.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Safety/bradycardia | 18 weeks
  We will evaluate for bradycardia after using the device at all time points using an EKG and heart rate variability (Beats/minute for each)

SECONDARY OUTCOMES:
Efficacy-cognition | initial visit, 2 weeks, 6 weeks, 12 weeks, 18 weeks
  We will assess whether vagus nerve simulation impacts clinical recovery from TBI as assessed by neuro-cognitive assessments
Efficacy-eye tracking | initial visit, 2 weeks, 6 weeks, 12 weeks, 18 weeks
  We will evaluate for changes in eye tracking metrics
Efficacy-serum biomarkers | initial visit, 2 weeks, 6 weeks, 12 weeks, 18 weeks
  Evaluate for changes in serum biomarkers with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Uzma Samadani, MD, PhD, Principal Investigator — Hennepin County Medical Center, Minneapolis; Thomas Bergman, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided